CLINICAL TRIAL: NCT02358187
Title: A Phase II Study of Vaccinations With HLA-A2 Restricted Glioma Antigen Peptides in Combination With Poly-ICLC for Children With Recurrent Unresectable Low-Grade Gliomas (LGG)
Brief Title: A Vaccine Trial for Low Grade Gliomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: James Felker (Other)
Collaborators: Connor's Cure (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, James Felker, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19060121; R01CA187219 (NIH); PRO13110086 (Other: Former identifier from University of Pittsburgh IRB)
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Low Grade Glioma
MeSH Terms: interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HLA-A2 Restricted Glioma Antigen-Peptides with Poly-ICLC (Experimental): All subjects will receive vaccine plus Poly-ICLC. Injections will be given every 3 week for a total of 8 vaccines.
  Interventions: Biological: Experimental: HLA-A2 Restricted Glioma Antigen-Peptides with Poly-ICLC

INTERVENTIONS:
Biological: Experimental: HLA-A2 Restricted Glioma Antigen-Peptides with Poly-ICLC — Poly-ICLC is administered intramuscularly (i.m.) using sterile technique, as supplied from the vial, and in the amount prescribed for the participant's weight. Patients should receive a dose of acetaminophen (15 mg/kg up to a max of 1000 mg) 30-60 minutes before each poly-ICLC administration. The poly-ICLC treatments will be administered immediately following the vaccine. Patients/parents will be asked to report any temperature elevations and side effects after each treatment.

SUMMARY:
The study will assess the immunogenicity, safety and preliminary clinical efficacy of the glioma associated antigen (GAA)/tetanus toxoid (TT) peptide vaccine and poly-ICLC in HLA-A2+ children with unresectable low-grade gliomas that have received at least two chemotherapy/biologic regimens. Radiation therapy counts as one biologic regimen, but patients may not have received radiation to the index lesion within 1 year of enrollment.

DETAILED DESCRIPTION:
Patients will be treated with subcutaneous injections of GAA/TT-vaccines starting on Week 0 and every 3 weeks thereafter for up to 8 cycles or until Off-treatment criteria are met (Section 4.6). I.m. poly-ICLC will be administered (30ug/kg i.m.) immediately following the vaccine. Poly-ICLC should be administered i.m. within 3 cm of the peptide-injection site.

To allow for flexibility with scheduling, the peptide vaccine and Poly-ICLC dose may be given within one week of the date that the vaccine and poly-ICLC administration are due.

Patients will be evaluated for any possible adverse event, regimen limiting toxicity (RLT) as well as clinical/radiological responses by clinical visits and MRI scanning. Follow-up MRIs will be performed (Weeks 6, 15 and 24).

ELIGIBILITY:
Inclusion Criteria:

Tumor Type

* Unresectable low-grade gliomas that have received at least two chemotherapy/biologic regimens. Radiation therapy counts as a biologic regimen. Patients may not have received radiation therapy to the index lesion within 1 year of enrollment. Patients may have tumor spread within the central nervous system (CNS).
* HLA-A2 positive based on flow cytometry.
* Patients must be clinically stable and off or on low-dose (no more than 0.1 mg/kg/day, max 4 mg/day Dexamethasone) corticosteroid for at least one week prior to study registration.
* Patients must be ≥ 12 months and < 22 years of age at the time of HLA-A2 screening.
* Patients must have a performance status of ≥ 70; (Karnofsky if > 16 years and Lansky if ≤ 16 years of age.
* Documented negative serum beta-human chorionic gonadotropin (HCG) for female patients who are post-menarchal. Because the effect of the peptide-based vaccine and poly-ICLC on the fetus has not sufficiently been investigated, pregnant females will not be included in the study.
* Patients must be free of systemic infection requiring IV antibiotics at the time of registration. Patients must be off IV antibiotics for at least 7 days prior to registration.
* Patients with adequate organ function as measured by: Bone marrow: absolute neutrophil count (ANC) > 1,000/µ; Platelets > 100,000/µ (transfusion independent); absolute lymphocyte count of ≥ 500/µ; Hemoglobin >8 g/dl (may be transfused). Hepatic: bilirubin < 1.5x institutional normal for age; serum glutamate pyruvate transaminase (SGPT) < 3x institutional normal.
* Renal: Serum creatinine based on age or Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70 ml/min/ml/min/1.73 m²
* Patients must have recovered from the toxic effects of prior therapy to grade 1 or better. Patients must be at least 3 weeks from the last dose of standard cytotoxic chemotherapy or myelosuppressive biological therapy and at least 1 week from the last dose of non-myelosuppressive biologic therapy.
* No overt cardiac, gastrointestinal, pulmonary or psychiatric disease.

Exclusion Criteria:

* Patients living outside of North America are not eligible.
* Patients may not have received radiation to the index lesion within 1 year of enrollment.
* Concurrent treatment or medications (must be off for at least 1 week) including:

  * Interferon (e.g. Intron-A®)
  * Allergy desensitization injections
  * Growth factors (e.g. Procrit®, Aranesp®, Neulasta®)
  * Interleukins (e.g. Proleukin®)
  * Any investigational therapeutic medication
* Patients must not have a history of, or currently active autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement.
* Use of immunosuppressives within four weeks prior to study entry or anticipated use of immunosuppressive agents. Dexamethasone, or other corticosteroid medications, if used in the peri-operative period must be tapered to no more than 0.1 mg/kg/day, max 4 mg/day dexamethasone for at least one week before study registration. Topical corticosteroids are acceptable.
* Because patients with immune deficiency are not expected to respond to this therapy, HIV-positive patients are excluded from the study.
* Patients who have received prior immunotherapy.

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-01; Primary Completion 2027-01-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor shrinkage or stable disease | Week 24
  Participants who demonstrate radiological evidence of tumor shrinkage or stable disease without regimen-limiting toxicity (RLT) after the initial 8 vaccines will be eligible to receive additional vaccinations beginning week 24 and every 6 weeks thereafter for up to two years.

CONTACTS AND LOCATIONS:
Overall Officials: James Felker, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States